CLINICAL TRIAL: NCT07309003
Title: Investigation of the Correlation With Clinical Data of the Effects of Functional Electrical Stimulation (FES) and Exercise on Quadriceps Muscle Strength and Structural Characteristics in Patients With Knee Osteoarthritis
Brief Title: The Effects of Functional Electrical Stimulation (FES) and Exercise on the Quadriceps in Patients With Knee Osteoarthritis
Status: Recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Betül KÜÇÜK GÜRSOY, DOCTOR, Ankara City Hospital Bilkent
Other Study IDs: TABED 2-24-28
Record Dates: First submitted 2025-11-18; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis (OA) of the Knee
Keywords: FES; Knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FES-Cycling: knee osteoarthritis
  Interventions: Device: functional electrical stimulation (FES)
- Cycling: knee osteoarthritis

INTERVENTIONS:
Device: functional electrical stimulation (FES) — FES-Cycling
  Groups: FES-Cycling

SUMMARY:
In our study, we aimed to compare the effects of functional electrical stimulation (FES) and an exercise program on quadriceps muscle strength and structural characteristics, as well as their impact on gait analysis, pain severity, and quality of life, in order to determine more effective and beneficial treatment programs for patients with knee OA.

DETAILED DESCRIPTION:
The study is planned as a prospective trial. Seventy patients, male or female, aged 50-65, who present to Ankara Bilkent City Hospital, Physical Therapy and Rehabilitation Hospital as outpatients, are diagnosed with osteoarthritis classified as Kellgren-Lawrence radiographic stage 2-3, and agree to participate in the study will be included.

According to the research criteria, initial evaluations will be conducted, and the demographic data (such as age, gender, height, weight, date of birth, occupation, systemic diseases) of eligible patients will be recorded by Dr. Betül Küçük Gürsoy. Patients' personal information will remain confidential and will not be shared with any person or institution/organization.

At the start of treatment, the VAS pain score, WOMAC, Quality of Life (SF-36) Scale, 6-Minute Walk Test (6-MWT), and Timed Up and Go Test (TUGT) will be recorded by Dr. Betül Küçük Gürsoy. Quadriceps muscle thickness and rectus femoris cross-sectional area will be measured via ultrasonography and recorded in a blinded manner by Dr. Ayşe Merve Ata.

Concurrently, isometric muscle strength measurements of the knee flexor and extensor groups using the Diers Myoline system will be performed and recorded in a blinded manner by Physiotherapist Selin Koç. Gait analysis (cadence, step length, stride length, step width, foot angle, and walking speed) using the Zebris FDM3 device will be conducted and recorded by Dr. Betül Küçük Gürsoy.

Subsequently, patients will be divided into two groups. The first group will receive aerobic exercise (stationary cycling) 5 times a week for a total of 10 sessions, administered by Dr. Betül Küçük Gürsoy. Additionally, they will be given a 6-week home exercise program to be performed 3 times a week, consisting of knee flexor and extensor range of motion exercises and isometric strengthening. The second group will receive Functional Electrical Stimulation-Cycling (FES-Cycling) 5 times a week for a total of 10 sessions, administered by Dr. Betül Küçük Gürsoy. They will also be given the same 6-week home exercise program (3 times a week) consisting of knee range of motion and isometric strengthening exercises.

ELIGIBILITY:
Inclusion Criteria:

* Being between 50-65 years of age
* Having knee OA (primary) according to ACR criteria
* Having grade 2-3 knee OA according to the Kellgren-Lawrence classification
* Having the ability to adhere to exercise regimens
* Agreeing to participate in the study

Exclusion Criteria:

* Having a diagnosis of secondary OA
* History of major knee trauma, surgery, or intra-articular steroid/hyaluronic acid injection in the last 6 months
* Presence of active synovitis
* Presence of neurological (Parkinson's, Alzheimer's, Polyneuropathy), endocrinological (diabetes mellitus), or vestibular disorders that could affect functional status, pain severity, or proprioception; or any disease that impairs these factors
* Pulmonary or cardiovascular disease that contraindicates exercise
* History of fracture and/or surgery in the lower extremity

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, male or female, aged 50-65, who present to Ankara Bilkent City Hospital Physical Therapy and Rehabilitation Hospital as outpatients, are diagnosed with osteoarthritis classified as Kellgren-Lawrence radiographic stage 2-3, and agree to participate in the study.
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Quadriceps muscle strength | From enrollment to the end of treatment at 6 weeks
  The patients' knee extensor and flexor muscle strengths were evaluated using the Diers Myoline Isometric Muscle Strength Measurement System. After positioning the individuals on the device, their name, surname, age, weight, and height information was recorded. They were then informed about how the test would be conducted and shown videos demonstrating the measurement procedure. For whichever muscle strength was being measured, they were instructed to perform the movement with maximal effort and to hold the muscle contraction isometrically for 10 seconds, after which the results were recorded.
  Measurement of patients' muscle strength before treatment, on the 10th day, and at the 6th week.
Visual Analog Scale (VAS) | From enrollment to the end of treatment at 6 weeks
  Zero indicates no pain at all, while 10 represents the worst possible pain.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara Bilkent Şehir Hastanesi, Ankara, Ankara
  - Ankara Bilkent City Hospital, Ankara

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Newham DJ, Donaldson Nde N. FES cycling. Acta Neurochir Suppl. 2007;97(Pt 1):395-402. doi: 10.1007/978-3-211-33079-1_52. PMID 17691402